CLINICAL TRIAL: NCT00639106
Title: The Use of Alloderm in Two-Stage, Tissue Expander/Implant Reconstruction: A Single-Blinded, Randomized, Controlled Trial
Brief Title: Tissue Expander/Implant Reconstruction: A Single-Blinded, Randomized, Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Michigan (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-024
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Breast expander; Breast reconstruction; implants; 08-024
MeSH Terms: conditions — Breast Neoplasms | interventions — Alloderm; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- A (Experimental): Expander Placement WITH Alloderm
  Interventions: Procedure: Alloderm, Questionnaires
- B (Active Comparator): Expander Placement WITHOUT Alloderm
  Interventions: Procedure: Without ALLODERM, Questionnaires

INTERVENTIONS:
Procedure: Alloderm, Questionnaires — All patients will undergo placement of a temporary tissue expander immediately following mastectomy.Patients will undergo the surgical creation of an expander pocket using implantable Alloderm.
  Other Names: Questionnaires administered prior to mastectomy, on Post-op Day #1, prior to the first, second; and third injection and following completion of expansion will take approximately 20 minutes; to complete.; It is expected that the panel of questionnaires administered at baseline (prior to mastectomy); and at 6 and 12 months following the exchange procedure will take approximately 45 minutes
  Arms: A
Procedure: Without ALLODERM, Questionnaires — A standard, sub-muscular pocket dissection will be performed in the patients assigned to the control group. No Alloderm will be used.
  Other Names: Questionnaires administered prior to mastectomy, on Post-op Day #1, prior to the first, second; and third injection and following completion of expansion will take approximately 20 minutes; to complete.; It is expected that the panel of questionnaires administered at baseline (prior to mastectomy); and at 6 and 12 months following the exchange procedure will take approximately 45 minutes
  Arms: B

SUMMARY:
Following mastectomy (removal of your breast), reconstruction of your breast(s) can be performed using tissue expanders and implants. At the same operation as your mastectomy, a tissue expander is put under the skin and muscles of your chest.

Following your surgery, the tissue expander is gradually filled with salt water over a period of months. Once the expander is filled to the size of your new breast, a second operation is performed. At this time, the tissue expander is removed and a permanent breast implant is placed. This is a standard procedure. We are interested in learning about the use of AlloDerm in breast reconstruction. AlloDerm can be used instead of some of your own chest muscles, in order to cover and protect a tissue expander. We want to know if the use of AlloDerm can decrease your pain or discomfort after surgery and after the filling of your tissue expander.

AlloDerm is made from human tissue. When AlloDerm is made all the cells that could cause your body to reject it are removed. When it is placed in your chest, your own cells will then grow into the AlloDerm, causing it to act like the muscle it is replacing. In this study, you will either have reconstruction with AlloDerm or without AlloDerm.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo immediate, postmastectomy, tissue expander/implant reconstruction
* Patients ≥ 21 and ≤ 75 years of age

Exclusion Criteria:

* Patient refusal
* Patients who will undergo any of the following:
* Single-stage implant reconstruction
* Combined autogenous tissue expander/implant reconstruction
* Patients with a history of prior irradiation
* Patients with a history of prior surgery with breast implants
* Patients with a history of prior axillary lymph node dissection
* Patients who are pregnant

The following eligibility will be confirmed at the time of surgery.

* Patients who are deemed intraoperatively by the attending surgeon to have significant mastectomy flap ischemia.
* Patients who have an axillary lymph node dissection at the time of mastectomy (Patients undergoing sentinel lymph biopsy are eligible)

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
whether using Alloderm to create the inferior-medial portion of the expander pocket will decrease patient-reported pain in both the immediate, post-operative period and during the expansion phase. | conclusion of the study

SECONDARY OUTCOMES:
To examine if the use of Alloderm will decrease patient-reported sensory morbidity in both the immediate, post-operative period and during the expansion phase. | conclusion of the study
To evaluate whether the use of Alloderm in tissue expander/implant reconstruction affects the rate of postoperative expansion and in-hospital narcotic use. | conclusion of the study
To examine if the use of Alloderm will impact both chronic breast pain and sensory morbidity. | conclusion of the study
To evaluate patient satisfaction following postmastectomy, tissue expander-implant reconstruction with and without the use of Alloderm. | conclusion of the study
To examine the effect of Alloderm on the overall aesthetic outcome, including the formation of capsular contracture, following tissue expander/implant reconstruction. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Disa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina

REFERENCES:
- [Derived] McCarthy CM, Lee CN, Halvorson EG, Riedel E, Pusic AL, Mehrara BJ, Disa JJ. The use of acellular dermal matrices in two-stage expander/implant reconstruction: a multicenter, blinded, randomized controlled trial. Plast Reconstr Surg. 2012 Nov;130(5 Suppl 2):57S-66S. doi: 10.1097/PRS.0b013e31825f05b4. PMID 23096987
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org